CLINICAL TRIAL: NCT06166498
Title: Effect of Single-course Malaria Chemoprevention on Clearance of and Protection From Plasmodium Falciparum Infection in the Presence of Resistance-associated Genotypes in Zambia
Brief Title: Parasite Clearance and Protection From Infection (PCPI) in Zambia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-KEP-813
Record Dates: First submitted 2023-11-29; First posted 2023-12-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-11

CONDITIONS: Malaria
Keywords: Malaria; Perennial malaria chemoprevention (PMC); Sulfadoxine-pyrimethamine (SP); Chemoprevention; Drug resistance
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate

STUDY DESIGN:
Intervention Model Description: Children assigned to group 1-SP will receive a 7-day course of placebo artesunate, whereas children in the group 2-AS will be given a 7-day course of active artesunate. This will span Day -7, -6, -5, -4, -3, -2, and -1. Then, on Day 0, children who had been given placebo artesunate will receive SP, whereas children in the AS group will receive placebo SP.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Fully placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulphadoxine-pyrimethamine (SP) (Active Comparator): Children in the SP group will receive a 7-day course of placebo artesunate (at day -7, -6, -5, -4, -3, -2, and -1), followed by the standard of care, 5 doses of SP.
  Interventions: Drug: SP (Macleods Pharmaceuticals Ltd)
- Artesunate monotherapy (AS) (Active Comparator): Children in the AS group will receive a 7-day course of 7-day course of active artesunate (at day -7, -6, -5, -4, -3, -2, and -1), followed by placebo SP.
  Interventions: Drug: AS (Guilin Pharmaceuticals)

INTERVENTIONS:
Drug: SP (Macleods Pharmaceuticals Ltd) — Children who weigh <10kg will receive Sulfadoxine-pyrimethamine paediatric formulation (250mg/12.5mg) dispersable tablets; children who weigh >10kg will receive 500mg sulfadoxine plus 25mg pyrimethamine
  Other Names: Sulfadoxine-pyrimethamine
  Arms: Sulphadoxine-pyrimethamine (SP)
Drug: AS (Guilin Pharmaceuticals) — Children will receive 4 mg/kg/day for 7 days
  Other Names: Artesunate
  Arms: Artesunate monotherapy (AS)

SUMMARY:
The Zambia PCPI study will measure the effect of the parasite genotypes associated with SP resistance on parasite clearance and protection from infection when exposed to SP. The total number of participants is expected to be 600 healthy between 3 to 5 years old who have no symptoms of malaria infection of which 400 children will be assigned to the SP group and 200 to the AS group. The results of this study will allow to measure the effect of the parasite genotypes associated with SP resistance on parasite clearance and protection from infection when exposed to SP.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recently published new malaria chemoprevention guidelines that included a recommendation for the provision of perennial malaria chemoprevention (PMC) with sulfadoxine-pyrimethamine (SP) to children resident in areas of high malaria transmission. PMC is the successor to an intervention originally known to as intermittent preventive treatment of malaria in infants (IPTi) that involved SP dosing of children at 2, 3 and 9 months of age during vaccination visits of the Essential Programme on Immunization (EPI) that coincide with the 2nd and 3rd doses of the DPT/Penta and measles vaccines. Under the new PMC guidelines, countries are now encouraged to increase the number and frequency of SP doses, and to extend the target age beyond the first year of life. Evidence supporting PMC comes in part from meta-analysis of six randomised placebo-controlled trials that demonstrated the protective effect of SP against clinical malaria, anaemia, hospital admissions due to malaria infection, and all-cause hospital admissions. Biomarkers of SP resistance, however, vary in different malaria-endemic settings and have been shown to compromise its protective effect.

In East and Southern Africa, Plasmodium falciparum parasites carry a high frequency of mutations in the Pfdhfr and Pfdhps genes with differing degrees of effect. In Mozambique, for example, SP was protective against malaria infection despite the Pfdhps A437G plus K540E double mutation circulating in over one-half, 52.3%, of P. falciparum (Pf) parasites.

In contrast, SP showed no protective effect in an IPTi trial in Northeastern Tanzania where 94.3% of Pf parasites had Pfdhps K540E. However, in this trial, the Pfdhps A581G mutation was also present in 55.0% of Pf parasites, forming the haplotype ISGEGA at codons 431, 436, 437, 540, 581 and 613. Thus, Pf appears to be highly resistant to SP where the A581G mutation is concurrently expressed with K540E. Fortunately, for PMC with SP there are few locations in East Africa where the combination of K540E and A581G circulate; most areas across Central, East and Southern Africa have parasites that contain the K540E without the A581G mutation (Pfdhps haplotype ISGEAA). The prevalence threshold of the ISGEAA haplotype at which SP is no longer protective is unknown. Indeed, there may not be an upper limit, although empirical studies are needed to confirm this.

In West Africa, specifically the Sahel region, there are emerging parasite genotypes that harbour a distinct haplotype of Pfdhps, VAGKGS, which lacks the K540E. These observations have come from molecular monitoring conducted alongside the delivery of intermittent preventive treatment of malaria in pregnancy (IPTp) with SP, and seasonal malaria chemoprevention (SMC) that targets children under 5 years of age with a combination of SP plus amodiaquine (AQ). The VAGKGS haplotype, and the related VAGKAS, have been reported in 2-40% of Pf parasites in Cameroon, Chad, Niger and Nigeria. The current distribution of parasites harbouring these genotypes is only partially described, and the effect these mutations have on parasite susceptibility to SP remains unknown. Nevertheless, it is possible that parasites harbouring Pfdhps-VAGKGS pose a threat to the effectiveness of PMC with SP or other SP-containing chemoprevention strategies in some parts of the West African Sahel. Thus, there are two clear evidence gaps, one in East/Southern Africa and another in West Africa, which the PCPI (parasite clearance and protection from infection) protocol has been developed to fill. This particular version of the PCPI protocol has been written for use in Zambia. Another PCPI protocol will be prepared for Cameroon with different sample sizes, but the approach will be the same.

The aim aim of this study is to evaluate a single-dose of malaria chemoprevention where genotypes (Pfdhps haplotypes ISGEAA and VAGKG/AS) are associated with SP resistance among healthy and symptom-free children between 3-5 years of age with unknown parasite status. In Zambia, the investigators objective is to measure parasite clearance and protection from infection conferred by malaria chemoprevention over a 63-day period in the presence/absence of the Pfdhps K540E mutation. In Cameroon, the objective will be to measure the same, but in the presence/absence of the VAGKGS haplotype.

The new WHO chemoprevention guidelines remove the upper age limit of 12 months so that countries may evaluate PMC among a broader range of ages. The investigators selected an age range for eligibility from 3 years and 0 days to 4 years and 364 days with the rationale being that 3-4 year olds are more likely to tolerate PMC dosing better than children 0-2 year olds. They are also more likely to have some modest level of semi-immunity and, therefore, are less likely to develop a clinical episode of malaria during the follow-up period relative to children who are 0-2 years of age.

After screening for eligibility, asymptomatic children based on a clinical examination and temperature reading will be randomised into one of two treatment groups on Day minus 7. Children randomised to the SP group will receive placebo artesunate monotherapy for seven consecutive days. On Day 0, these children will then be given SP. In contrast, children randomised into the AS group will receive active artesunate monotherapy for seven consecutive days and then SP placebo on Day 0. The AS group will establish one sub-set of children who are parasite-free at Day 0, and allow for an accurate estimate of background incidence (reflecting transmission intensity) to which all groups will be exposed during follow up. In addition, this group allows a more accurate estimation of underlying frequency of Pfdhps 540E mutations in the parasite population. Part of the rationale, as well, is to look at parasite clearance among those who were qPCR-positive at Day 0 and time to incident infection among qPCR-negative at Day 0. This will inform parameters of models the investigators will use in data analyses. All will be followed 70 days total, 63 days (9-week period total) following treatment.

Summary of treatments and children per group Treatment sulfadoxine-pyrimethamine (SP)* artesunate monotherapy (AS)**

*Seven-day course of daily placebo artesunate to be included starting on Day -7

**Seven-day course of artesunate beginning on Day -7 followed by a single-course of SP placebo at Day 0

Sample collection will be conducted at scheduled visits on Days 0, 2, 5, 7, 14, 21, and 28 visits as children provide a pin-prick of blood for a film slide and a dried blood-spot (DBS) on filter paper. On Days 35, 42, 49, 56, and 63 visits, only DBS will be collected. A study physician will be available 24 hours a day for unscheduled visits to review study subjects who develop symptoms.

All children will be screened for malaria symptoms, including a temperature check, at all contacts - scheduled visits and unscheduled visits - during their involvement in the study. All symptomatic children will have a malaria rapid diagnostic test (RDT) administered and a blood film taken. If a child is RDT-positive at any scheduled or unscheduled visit, the RDT will be stored for future genotyping rather than collecting a separate DBS. In all instances of a positive RDT, children will receive a full course of first-line therapy, artemether-lumefantrine (AL). Children who have an RDT diagnosis will no longer contribute to any future endpoints of the trial, but they will be asked to continue with symptom screening for the full follow-up period to Day 63 and, if symptomatic, they will be tested by RDT and again treated with first-line therapy if found positive and at least 28 days have elapsed since their previous AL-treated febrile episode. Where a child has a second febrile episode within 28 days with RDT-confirmed recurrent parasitaemia, the second-line treatment in Zambia, dihydroartemisinin-piperaquine (DP), will be administered. This ensures quality care is equitable for all participants, regardless of treatment group allocation.

The duration of follow-up in the PCPI protocol was carefully considered. Most study designs of malaria treatment efficacy have a primary endpoint of parasitaemia (present/absent) measured by slide microscopy at Day 28 (4 weeks) with PCR correction, an approach also outlined in the new WHO chemoprevention efficacy study (CPES) protocol. This study is consistent with procedures for the PCPI protocol. Consequently, data derived from PCPI studies will be comparable with data from other studies, including those conducted using the CPES protocol. The CPES protocol defines chemoprevention efficacy as both the ability to clear existing parasites and prevent a new infection for a short period (of 28 days). However, PCPI studies will separate resistance effects on these two outcomes of clearance and protection and extend the follow up period to Day 63 (9 weeks). This allows for better quantification of the protective efficacy against new infections by genotype, particularly when the mean duration of protection against more sensitive strains is higher or close to 28 days. Additionally, the choice of a 63-day follow-up simulates what might be the protective efficacy in a scenario where chemoprevention is administered to children every two months. This will be increasingly important for comparison purposes through meta-analyses as longer-acting interventions, including introduction of monoclonal therapies and malaria vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Be 3-5 years old
* Exhibit no symptoms of malaria
* Have parents/guardians willing to have their child participate in all follow-up visits and seek care from study staff
* Reside in the study catchment area

Exclusion Criteria:

* Have evidence of acute illness as determined by clinical examination
* Exhibit symptoms of malaria (axillary fever ≥ 37.5 °C and / or history of fever in past 48 hours)
* Have known allergy to study medications
* Have received antimalarial treatment or azithromycin within 28 days prior to screening
* Be concomitantly receiving co-trimoxazole (trimethoprim-sulfamethoxazole)
* Be categorised as severely malnourished according to WHO child growth standards

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Parasite clearance | 28 days (total follow up 63 days post SP dose)
  Time to clearance of parasite genotypes among SP recipients who were positive on Day 0 by qPCR presence/absence of Pfdhps K540E and measured to Day 63
Protection from infection | 28 days (total follow up 63 days post SP dose)
  (a) Mean duration of SP protection against parasite genotypes determined by Pfdhps gene sequence presence/absence of Pfdhps K540E among SP recipients who were parasite-free on Day 0 by qPCR (b) Mean duration of symptom-free status among SP recipients who were parasite free on Day 0 by qPCR, stratified by parasite Pfdhps genotype at time of febrile malaria episode

SECONDARY OUTCOMES:
Parasite clearance | 7 days (day -7 until day 0)
  Time to clearance of parasite genotypes among AS recipients positive at Day -7 by qPCR (presence/absence of Pfdhps K540E) and measured to Day 0
Protection from infection | Time Frame: 35 days (day 0 until day 35)
  (a) Mean duration of AS protection by qPCR (b) Mean duration of symptom-free status among AS recipients

CONTACTS AND LOCATIONS:
Overall Officials: R Matthew Chico, MPH, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Nchelenge District, Nchelenge, Luapula Province, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. WHO guidelines for malaria, 3 June 2022: World Health Organization, 2022.
- [Background] Aponte JJ, Schellenberg D, Egan A, Breckenridge A, Carneiro I, Critchley J, Danquah I, Dodoo A, Kobbe R, Lell B, May J, Premji Z, Sanz S, Sevene E, Soulaymani-Becheikh R, Winstanley P, Adjei S, Anemana S, Chandramohan D, Issifou S, Mockenhaupt F, Owusu-Agyei S, Greenwood B, Grobusch MP, Kremsner PG, Macete E, Mshinda H, Newman RD, Slutsker L, Tanner M, Alonso P, Menendez C. Efficacy and safety of intermittent preventive treatment with sulfadoxine-pyrimethamine for malaria in African infants: a pooled analysis of six randomised, placebo-controlled trials. Lancet. 2009 Oct 31;374(9700):1533-42. doi: 10.1016/S0140-6736(09)61258-7. Epub 2009 Sep 16. PMID 19765816
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Chandramohan D, Owusu-Agyei S, Carneiro I, Awine T, Amponsa-Achiano K, Mensah N, Jaffar S, Baiden R, Hodgson A, Binka F, Greenwood B. Cluster randomised trial of intermittent preventive treatment for malaria in infants in area of high, seasonal transmission in Ghana. BMJ. 2005 Oct 1;331(7519):727-33. doi: 10.1136/bmj.331.7519.727. PMID 16195288
- [Background] Macete E, Aide P, Aponte JJ, Sanz S, Mandomando I, Espasa M, Sigauque B, Dobano C, Mabunda S, DgeDge M, Alonso P, Menendez C. Intermittent preventive treatment for malaria control administered at the time of routine vaccinations in Mozambican infants: a randomized, placebo-controlled trial. J Infect Dis. 2006 Aug 1;194(3):276-85. doi: 10.1086/505431. Epub 2006 Jun 30. PMID 16826474
- [Background] Kobbe R, Kreuzberg C, Adjei S, Thompson B, Langefeld I, Thompson PA, Abruquah HH, Kreuels B, Ayim M, Busch W, Marks F, Amoah K, Opoku E, Meyer CG, Adjei O, May J. A randomized controlled trial of extended intermittent preventive antimalarial treatment in infants. Clin Infect Dis. 2007 Jul 1;45(1):16-25. doi: 10.1086/518575. Epub 2007 May 29. PMID 17554695
- [Background] Mockenhaupt FP, Reither K, Zanger P, Roepcke F, Danquah I, Saad E, Ziniel P, Dzisi SY, Frempong M, Agana-Nsiire P, Amoo-Sakyi F, Otchwemah R, Cramer JP, Anemana SD, Dietz E, Bienzle U. Intermittent preventive treatment in infants as a means of malaria control: a randomized, double-blind, placebo-controlled trial in northern Ghana. Antimicrob Agents Chemother. 2007 Sep;51(9):3273-81. doi: 10.1128/AAC.00513-07. Epub 2007 Jul 16. PMID 17638703
- [Background] Grobusch MP, Lell B, Schwarz NG, Gabor J, Dornemann J, Potschke M, Oyakhirome S, Kiessling GC, Necek M, Langin MU, Klein Klouwenberg P, Klopfer A, Naumann B, Altun H, Agnandji ST, Goesch J, Decker M, Salazar CL, Supan C, Kombila DU, Borchert L, Koster KB, Pongratz P, Adegnika AA, Glasenapp Iv, Issifou S, Kremsner PG. Intermittent preventive treatment against malaria in infants in Gabon--a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2007 Dec 1;196(11):1595-602. doi: 10.1086/522160. Epub 2007 Oct 25. PMID 18008242
- [Background] Mayor A, Serra-Casas E, Sanz S, Aponte JJ, Macete E, Mandomando I, Puyol L, Berzosa P, Dobano C, Aide P, Sacarlal J, Benito A, Alonso P, Menendez C. Molecular markers of resistance to sulfadoxine-pyrimethamine during intermittent preventive treatment for malaria in Mozambican infants. J Infect Dis. 2008 Jun 15;197(12):1737-42. doi: 10.1086/588144. PMID 18419347
- [Background] Gupta H, Macete E, Bulo H, Salvador C, Warsame M, Carvalho E, Menard D, Ringwald P, Bassat Q, Enosse S, Mayor A. Drug-Resistant Polymorphisms and Copy Numbers in Plasmodium falciparum, Mozambique, 2015. Emerg Infect Dis. 2018 Jan;24(1):40-48. doi: 10.3201/eid2401.170864. PMID 29260689
- [Background] Gosling RD, Gesase S, Mosha JF, Carneiro I, Hashim R, Lemnge M, Mosha FW, Greenwood B, Chandramohan D. Protective efficacy and safety of three antimalarial regimens for intermittent preventive treatment for malaria in infants: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Oct 31;374(9700):1521-32. doi: 10.1016/S0140-6736(09)60997-1. Epub 2009 Sep 16. PMID 19765815
- [Background] Naidoo I, Roper C. Mapping 'partially resistant', 'fully resistant', and 'super resistant' malaria. Trends Parasitol. 2013 Oct;29(10):505-15. doi: 10.1016/j.pt.2013.08.002. Epub 2013 Sep 9. PMID 24028889
- [Background] Oguike MC, Falade CO, Shu E, Enato IG, Watila I, Baba ES, Bruce J, Webster J, Hamade P, Meek S, Chandramohan D, Sutherland CJ, Warhurst D, Roper C. Molecular determinants of sulfadoxine-pyrimethamine resistance in Plasmodium falciparum in Nigeria and the regional emergence of dhps 431V. Int J Parasitol Drugs Drug Resist. 2016 Dec;6(3):220-229. doi: 10.1016/j.ijpddr.2016.08.004. Epub 2016 Sep 29. PMID 27821281
- [Background] ACCESS-SMC Partnership. Effectiveness of seasonal malaria chemoprevention at scale in west and central Africa: an observational study. Lancet. 2020 Dec 5;396(10265):1829-1840. doi: 10.1016/S0140-6736(20)32227-3. PMID 33278936
- [Background] World Health Organisation. Malaria chemoprevention efficacy study protocol. Geneva: World Health Organisation, 2022.
- [Derived] Martinez-Vega R, Chaponda M, Mousa A, Gwasupika J, Chaponda EB, Daka V, Mwanza S, Chipunga M, Beshir KB, Chopo-Pizarro A, Kaur H, Okell L, Hansson H, Hocke EF, Alifrangis M, Gosling R, Roper C, Sutherland C, Chico RM. Parasite clearance and protection from Plasmodium falciparum infection (PCPI): a two-arm, parallel, double-blinded, placebo-controlled, randomised trial of presumptive sulfadoxine-pyrimethamine versus artesunate monotherapy among asymptomatic children 3-5 years of age in Zambia. BMC Infect Dis. 2025 Nov 11;25(1):1547. doi: 10.1186/s12879-025-11975-3. PMID 41219832